CLINICAL TRIAL: NCT01310309
Title: EXecutive Registry: XIENCE V® Everolimus Eluting Coronary Stent System (XIENCE V® EECSS) in the Treatment of the Specific Setting of Patients With Multi-vessel Coronary Artery Disease.
Brief Title: EXecutive Registry: Evaluating XIENCE V® in a Multi Vessel Disease
Acronym: EXecutive
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 07-380 Registry
Record Dates: First submitted 2011-03-03; First posted 2011-03-08 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: Coronary Disease; Coronary Artery Disease; Coronary Artery Stenosis; Coronary Artery Restenosis
Keywords: Stents; Drug-eluting Stent; Angioplasty; Coronary Artery stenosis; Coronary Artery Stent Restenosis; Stent Thrombosis
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease; Coronary Stenosis; Coronary Restenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- EXecutive Registry: A prospective controlled registry to analyze the clinical efficacy and safety at mid and long-term follow-up in patients with MVD treated with the XIENCE V® Everolimus Eluting Coronary Stent System (XIENCE V® EECSS).
  Interventions: Device: Coronary artery placement of a drug-eluting stent

INTERVENTIONS:
Device: Coronary artery placement of a drug-eluting stent — Coronary artery placement of a drug-eluting stent (XIENCE V® EECSS)

SUMMARY:
The purpose of this two part study is the assessment of the performance of the XIENCE V® Everolimus Eluting Coronary Stent System (XIENCE V® EECSS) in the treatment of the specific setting of patients with Multi-Vessel Coronary Artery Disease (MVD).

DETAILED DESCRIPTION:
This is a clinical evaluation of the XIENCE V® everolimus eluting coronary stent system as a revascularization treatment of patients with multi-vessel coronary artery disease (MVD-CAD).

The sutdy is composed of two parts:

A Randomized Controlled Trial, outlined in a separate posting and the registry portion of this study, which is as follows:

-A prospective controlled registry to analyze the clinical efficacy and safety at mid and long-term follow-up in patients with MVD treated with the XIENCE V® Everolimus Eluting Coronary Stent System (XIENCE V® EECSS).

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be at least 18 years of age
2. Patient is able to verbally confirm understanding of risks, benefits and treatment alternatives of receiving the XIENCE V® EECSS and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure, as approved by the appropriate Medical Ethics Committee of the respective clinical site
3. Patient has been diagnosed a MVD, as documented by coronary angiography, i.e. presenting a severe stenosis (>50%) amenable to PCI in at least 2 major epicardial vessels or their principal bifurcation branches (diagonal or obtuse marginal)
4. Patient must have evidence of myocardial ischemia (e.g., stable or unstable angina, silent ischemia, positive functional study or a reversible change in the electrocardiogram -ECG- consistent with ischemia)
5. Patient must be an acceptable candidate for coronary artery bypass graft (CABG) surgery
6. Patient must agree to undergo all protocol-required follow-up examinations.

Angiographic Inclusion Criteria

1. Patients may receive up to 4 planned XIENCE V® EECSS stents, depending on the number of vessels treated and their respective lesion length. When multiple lesions are present in one or more main coronary branches, complete revascularization should be attempted with the implantation of a maximum of 4 planned stents
2. Target lesions must be de novo lesions (no prior stent implant, no prior brachytherapy)
3. Target vessel reference diameter must be between 2.5 mm and 4.0 mm by visual estimate
4. Target lesion < or = 28 mm in length by visual estimation
5. Target lesions must be in a major artery or its principal branches (diagonal or obtuse marginal) with a visually estimated stenosis of > or = 50%
6. Two lesions in a single main coronary artery or its branches do not constitute a MVD situation, therefore this type of patient must not be enrolled

Exclusion Criteria:

1. Patient has had a known diagnosis of acute myocardial infarction (AMI) within 72 hours preceding the index procedure (non-procedural/spontaneous MI, CK-MB > or = to 2 times upper limit of normal) and CK and CK-MB have not returned within normal limits at the time of procedure
2. Patient has current unstable arrhythmias
3. Patient has a known left ventricular ejection fraction (LVEF) <30%
4. Patient has received a heart transplant or any other organ transplant or is on a waiting list for any organ transplant
5. Patient is receiving or scheduled to receive chemotherapy or radiation therapy within 30 days prior to or after the procedure.
6. Patient is receiving immunosuppression therapy or has known immunosuppressive or autoimmune disease (e.g. human immunodeficiency virus, systemic lupus erythematosus etc.)
7. Patient is receiving chronic anticoagulation therapy (e.g. coumadin)
8. Patient has a known hypersensitivity or contraindication to aspirin, paclitaxel, either heparin or bivalirudin, clopidogrel or ticlopidine, everolimus, cobalt, chromium, nickel, tungsten, acrylic and fluoro polymers or contrast sensitivity that cannot be adequately pre-medicated
9. Elective surgery is planned within the first 9 months (+/- 14 days) after the procedure that will require discontinuing either aspirin or clopidogrel
10. Patient has a platelet count <100,000 cells/mm3 or >700,000 cells/mm3, a WBC of <3,000 cells/mm3, or documented or suspected liver disease (including laboratory evidence of hepatitis)
11. Patient has known renal insufficiency (e.g., serum creatinine level of more than 2.5 mg/dl, patient on dialysis)
12. Patient has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions
13. Patient has had a cerebrovascular accident (CVA) or transient ischemic neurological attack (TIA) within the past six months
14. Patient has had a significant GI or urinary bleed within the past six months
15. Patient has other medical illness (e.g., cancer or congestive heart failure) or known history of substance abuse (alcohol, cocaine, heroin etc.) that may cause non-compliance with the protocol, confound the data interpretation or is associated with a limited life expectancy (i.e. less than one year)
16. Patient is already participating in another investigational use device or drug study or has completed the follow-up phase of another study within the last 30 days.

Angiographic Exclusion Criteria

1. Target lesion meets any of the following criteria:

   * Left main location
   * Located within an arterial or saphenous vein graft or distal to a diseased arterial or saphenous vein graft (defined as vessel irregularity per angiogram and >20% stenosed lesion by visual estimation)
   * Heavy calcification
2. The patient may need more than 4 planned stents. Bailout stents are allowed but must be of the same type as randomization stent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Multi-Vessel Coronary Artery Disease (MVD) treated with the XIENCE V® Everolimus Eluting Coronary Stent System (XIENCE V® EECSS).
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2007-09; Primary Completion 2010-10 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Composite endpoint of all Death, MI (Q-wave and non Q-wave), and ischemia-driven Target Vessel Revascularization (TVR) . | 12 months
  Composite endpoints are endpoints made up of a range of statistical parameters.

SECONDARY OUTCOMES:
Adjudicated stent thrombosis | 30 days
Revascularizations (TLR/TVR/any revascularization) | 30 days
Composite endpoint of cardiac death, MI (Q-wave and non Q-wave), and ischemia-driven TLR. | 30 days
Composite endpoint of all death, MI (Q-wave and non Q-wave), and TVR. | 30 days
Device success | At time of index procedure
  Achievement of a final residual in-stent diameter stenosis of < 30% (visual assessment) using the assigned device only.
Lesion success | At time of index procedure
  Attainment of < 30% residual in-stent stenosis (by visual assessment) using any percutaneous method.
Procedural success defined as: residual in-stent %DS of < 30% using a percutaneous method, without cardiac death, Q-wave MI, non Q-wave MI, or repeat revasc of the target during hospitalization. | At time of index procedure
Adjudicated stent thrombosis | 1 year
Adjudicated stent thrombosis | 2 years
Adjudicated stent thrombosis | at 3 years
Revascularizations (TLR/TVR/any revascularization) | 1 year
Revascularizations (TLR/TVR/any revascularization) | 2 years
Revascularizations (TLR/TVR/any revascularization) | 3 years
Composite endpoint of cardiac death, MI (Q-wave and non Q-wave), and ischemia-driven TLR. | 1 years
Composite endpoint of cardiac death, MI (Q-wave and non Q-wave), and ischemia-driven TLR. | 2 years
Composite endpoint of cardiac death, MI (Q-wave and non Q-wave), and ischemia-driven TLR. | 3 years
Composite endpoint of all death, MI (Q-wave and non Q-wave), and TVR. | 2 years
Composite endpoint of all death, MI (Q-wave and non Q-wave), and TVR. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Corrado Vassanelli, MD, Principal Investigator — Ospedale Civile Maggiore - Università di Verona; Flavio Ribichini, MD, Principal Investigator — Ospedale Civile Maggiore - Università di Verona
Locations (23):
- Italy (23):
  - A.O. San Giovanni di Dio, Agrigento
  - Ospedale Maggiore Bologna, Bologna
  - Policlinico S. Orsola - Malpighi, Bologna
  - A.O. Cannizzaro, Catania
  - A.O. Universitaria Vittorio Emanuele - Ferrarotto - S. Bambino, Catania
  - A.O. Università Mater Domini c/o Campus Università Magna Grecia, Catanzaro
  - A.O. Universitaria OO.RR Foggia, Foggia
  - E.O. Ospedali Galliera, Genova
  - A.O. Carlo Poma, Mantova
  - Centro Cardiologico Monzino, Milan
  - Ospedale Loreto Mare, Napoli
  - A. O. Sant'Andrea, Roma
  - Ospedale Generale Madre Vannini, Roma
  - Ospedale Sandro Pertini, Roma
  - A.S.O. Molinette San Giovanni Battista di Torino, Torino
  - Ospedale Maria Vittoria, Torino
  - P.O. San Giovanni Bosco, Torino
  - San Giovanni Battista - Ospedale Molinette, Torino
  - A.O. Universitaria - Ospedale Riuniti Umberto I - G.M. Lancisi - G. Salesi, Torrette Di Ancona
  - Ospedale Civile Maggiore - Università di Verona, Verona
  - Ospedale Civile, Vicenza
  - Ospedale Civile di Vigevano, Vigevano
  - A.O. Della Provincia di Pavia, Voghera